CLINICAL TRIAL: NCT04873934
Title: A Randomized, Controlled, Multicenter, Open-label Trial Comparing a Hospital Post-discharge Care Pathway Involving Aggressive LDL-C Management That Includes Inclisiran With Usual Care Versus Usual Care Alone in Patients With a Recent Acute Coronary Syndrome (VICTORION-INCEPTION)
Brief Title: Management of LDL-cholesterol With Inclisiran + Usual Care Compared to Usual Care Alone in Participants With a Recent Acute Coronary Syndrome
Acronym: V-INCEPTION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CKJX839A1US01
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Results first posted 2025-08-21 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Acute Coronary Syndrome
Keywords: Hyperlipidemia; Atherosclerotic Cardiovascular Disease; Hypercholesterolemia; Lipid lowering therapies
MeSH Terms: conditions — Acute Coronary Syndrome; Hyperlipidemias; Atherosclerosis; Hypercholesterolemia | interventions — ALN-PCS

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inclisiran with Usual Care (Experimental): Inclisiran sodium 300 mg / 1.5 ml (equivalent to 284 mg of inclisiran)
  Interventions: Drug: Inclisiran
- Usual Care (No Intervention): Usual Care Alone

INTERVENTIONS:
Drug: Inclisiran — Inclisiran sodium 300 mg / 1.5 ml (equivalent to 284 mg of inclisiran)
  Other Names: KJX839
  Arms: Inclisiran with Usual Care

SUMMARY:
The purpose of this study is to study the effectiveness of implementation of a systematic LDL-C management pathway including treatment with inclisiran in participants who have experienced a recent acute coronary syndrome (ACS) and have an increased LDL-cholesterol (≥70 mg/dL) despite being treated with a statin drug.

DETAILED DESCRIPTION:
This was a randomized, parallel-group, open-label, multicenter, 1-year (30-day Screening Period and 330-day Treatment Period) study comparing an LDL-C management strategy including inclisiran + usual care to usual care alone. Approximately 384 participants were planned to be randomized 1:1 to aggressive LDL-C management with inclisiran + usual care (intervention arm) (3 inclisiran doses) or usual care (control arm). Usual care could have included addition of ezetimibe, bempedoic acid, PCSK9-inhibiting monoclonal antibodies, and/or commercially available inclisiran

ELIGIBILITY:
Inclusion Criteria:

* Recent Acute Coronary Syndrome (in-patient/out-patient) within 5 weeks of screening
* Serum LDL-C ≥70 mg/dL or non-HDL-C ≥100 mg/dL
* Fasting triglycerides <4.52 mmol/L (<400 mg/dL) at screening
* Calculated glomerular filtration rate >20 mL/min by estimated glomerular filtration rate (eGFR)
* Participants are required to be discharged on statin therapy, or have documented statin intolerance, as determined by the investigator, following hospitalization for an ACS. Statin intolerant participants are eligible if they had intolerable side effects on at least 2 different statins, including one at the lowest standard dose

Exclusion Criteria:

* New York Heart Association (NYHA) class IIIb or IV heart failure or last known left ventricular ejection fraction <25%.
* Significant cardiac arrhythmia within 3 months prior to randomization that is not controlled by medication or via ablation at the time of screening.
* Severe concomitant non-cardiovascular disease that carries the risk of reducing life expectancy to less than 2 years.
* Treatment with other investigational products or devices within 30 days or five half˗lives of the screening visit, whichever is longer.
* Planned use of other investigational products or devices during the course of the study.
* Treatment with monoclonal antibodies directed towards PCSK9 within 90 days of screening.
* Recurrent ACS event within 2 weeks prior to randomization.
* Coronary angiography and revascularization procedure (percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG) surgery) performed within 2 weeks prior to the randomization visit or planned after randomization.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2024-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (88):
- United States (88):
  - Northeast Arkansas Baptist Clinic, Jonesboro, Arkansas
  - Central Cardiology Medical Center, Bakersfield, California
  - The Heart Group Cardiovascular Associates Inc, Fresno, California
  - Mission Heritage Medical Group, Mission Viejo, California
  - Northbay Clinical Research LLC, Santa Rosa, California
  - Clinnova Research Solutions, Torrance, California
  - Harbor-UCLA Medical Center, Torrance, California
  - Interv Cardiology Med Grp, West Hills, California
  - Aurora Denver Cardiology Associates, Aurora, Colorado
  - Colorado Springs Cardiology, Colorado Springs, Colorado
  - Colorado Heart and Vascular, Lakewood, Colorado
  - Cardiology Ass of Fairfield County, Stamford, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - George Washington Univ Medical Ctr, Washington D.C., District of Columbia
  - Nova Clinical Research LLC, Bradenton, Florida
  - Teradan Clinical trials LLC, Brandon, Florida
  - Clearwater Cardiovascular and Interventional Consultants, Clearwater, Florida
  - Cardiology Research Associates, Daytona Beach, Florida
  - Holy Cross Hospital Inc, Fort Lauderdale, Florida
  - Baptist Health Research Institute, Jacksonville, Florida
  - Reliant Medical Research, Miami, Florida
  - Inpatient Research Clinical LLC, Miami Lakes, Florida
  - Innovation Medical Group LLC, Palmetto Bay, Florida
  - Cardiology Consultants, Pensacola, Florida
  - Theia Clinical Research Ctrs LLC, Tampa, Florida
  - Morehouse School Of Medicine, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Ellipsis Group, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northwest Heart Clinical Rsrch LLC, Arlington Heights, Illinois
  - AMITA Heart and Vascular Group, Hinsdale, Illinois
  - Franciscan Health Services Research Center, Indianapolis, Indiana
  - Cardiovascular Research Of Northwest Indiana, Llc, Munster, Indiana
  - Iowa Heart Center, Des Moines, Iowa
  - Midwest Heart and Vascular Spec, Overland Park, Kansas
  - Tidal Health Peninsula Regional Inc, Salisbury, Maryland
  - Sparrow Clincal Research Institute, Lansing, Michigan
  - MidMichigan Physicians Group, Midland, Michigan
  - St Marys of Ascension Research, Saginaw, Michigan
  - Trinity Health Michigan Heart, Ypsilanti, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - CentraCare Heart and Vascular Center, Saint Cloud, Minnesota
  - Jackson Heart Clinic, Jackson, Mississippi
  - Cardiology Associates of North MS, Tupelo, Mississippi
  - St Louis Heart and Vascular, St Louis, Missouri
  - Bryan LGH Heart Inst Intigrated Cardiology Group, Lincoln, Nebraska
  - Meridian Clinical Research, Lincoln, Nebraska
  - Advanced Heart Care, LLC, Bridgewater, New Jersey
  - Cardiovas Assoc of Delaware Valley, Elmer, New Jersey
  - Inspira Medical Cent Mullica Hill, Mullica Hill, New Jersey
  - Capital Cardiology Associates, Albany, New York
  - University At Buffalo, Buffalo, New York
  - Bassett Medical Center, Cooperstown, New York
  - Jamaica Hospital Medical Center, Jamaica, New York
  - Northwell Health, Manhasset, New York
  - Laurelton Heart Specialist PC, Rosedale, New York
  - Cary Research Group, Cary, North Carolina
  - Moses Cone Hospital-Lebauer CV Research Foundation, Greensboro, North Carolina
  - Clinical Trials Of America LLC, Lenoir, North Carolina
  - Pinehurst Medical Clinic, Pinehurst, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Aultman Hospital, Canton, Ohio
  - University of Toledo, Toledo, Ohio
  - St John Health System, Bartlesville, Oklahoma
  - Bend Memorial Clinic, Bend, Oregon
  - University of Pittsburgh Medical Center HABOT, Erie, Pennsylvania
  - Lancaster General Health, Lancaster, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Guthrie Clinic, Sayre, Pennsylvania
  - Monument Health Clinical Research, Rapid City, South Dakota
  - Covenant Medical Group, Knoxville, Tennessee
  - Baylor Scott and White Heart and Vascular Hospital, Dallas, Texas
  - Vilo Research Group LLC, Houston, Texas
  - Texas Heart Medical Group, Houston, Texas
  - UT Physicians Memorial Hermann, Houston, Texas
  - Northwest Houston Cardiology PA, Houston, Texas
  - West Houston Area Clinical Trial Consultants, Houston, Texas
  - The Heart Institute of East Texas, Lufkin, Texas
  - CardioVoyage LLC, McKinney, Texas
  - Research Group of North Texas, Sunnyvale, Texas
  - Tyler Cardiovascular Consultants, Tyler, Texas
  - Intermountain Medical Center, Murray, Utah
  - TPMG Clinical Research, Newport News, Virginia
  - York Clinical Research, Norfolk, Virginia
  - Dominion Medical Associates, Richmond, Virginia
  - Carilion Clinic, Roanoke, Virginia
  - Selma Medical Associates, Winchester, Virginia
  - MultiCare Institute for Research and Innovation, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2749

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 87 study centers. Of the 201 participants randomized to inclisiran + usual care, 1 participant was randomized erroneously and did not receive inclisiran. Of the 199 participants randomized to usual care, 3 participants received commercially available inclisiran as part of their concomitant medications.
Groups:
- Inclisiran With Usual Care: Inclisiran sodium 300 mg / 1.5 ml (equivalent to 284 mg of inclisiran) + usual care
Period: Overall Study
Arm/Group | Inclisiran With Usual Care | Usual Care
Started | 201 | 199
Full Analysis Set (Full Analysis Set (FAS) included all randomized participants) | 201 | 199
Safety Set (Safety Set included all participants who received study treatment. Participants in the usual care treatment group who had data collected at the baseline visit were included in the Safety Set.) | 203 | 197
Completed | 183 | 173
Not Completed | 18 | 26
Not completed — Adverse Event | 0 | 1
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 13 | 9
Not completed — Physician Decision | 1 | 1
Not completed — Protocol deviation | 2 | 1
Not completed — Subject decision | 1 | 8
Not completed — Withdrew consent | 0 | 4
Not completed — Missing | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inclisiran With Usual Care | Usual Care | Total
Number analyzed (Participants) | 201 | 199 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (10.90) | 60.2 (11.69) | 60.5 (11.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 53 | 116
  Male | 138 | 146 | 284
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 166 | 167 | 333
  Black or African American | 25 | 24 | 49
  Asian | 6 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  American Indian or Alaska Native | 1 | 0 | 1
  Unknown | 2 | 4 | 6
  Multiple | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Day 330 in LDL-C
Description: Percent change from baseline in Low-Density Lipoprotein Cholesterol (LDL-C) at Day 330
Time Frame: Baseline and Day 330
Population: Full Analysis Set (FAS) comprised all randomized participants. The number of participants analyzed corresponds to the number of subjects who had LDL-C values at baseline and Day 330.
Measure: Least Squares Mean (97.5% Confidence Interval); unit: Percent change in LDL-C
Arm/Group | Inclisiran With Usual Care | Usual Care
Number analyzed (Participants) | 171 | 163
Percent change in LDL-C | -45.6 [-51.5 to -39.6] | 1.4 [-4.7 to 7.5]
Statistical Analysis 1: Comparison: Inclisiran With Usual Care vs Usual Care; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS mean difference = -46.9, 97.5% CI 2-sided [-55.4 to -38.5]

2. Primary Outcome: Achievement of LDL-C < 70 mg/dL at Day 330
Description: Percentage of participants achieving Low-Density Lipoprotein Cholesterol (LDL-C) < 70 mg/dL at Day 330
Time Frame: Day 330
Population: Full Analysis Set (FAS) comprised all randomized participants.
Measure: Number (97.5% Confidence Interval); unit: Percentage of participants
Arm/Group | Inclisiran With Usual Care | Usual Care
Number analyzed (Participants) | 201 | 199
Percentage of participants | 66.7 [59.2 to 74.1] | 28.1 [21.0 to 35.3]
Statistical Analysis 1: Comparison: Inclisiran With Usual Care vs Usual Care; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 5.42, 97.5% CI 2-sided [3.29 to 8.91]

3. Secondary Outcome: Absolute Change From Baseline in LDL-C
Description: Absolute change from baseline in low-density lipoprotein cholesterol (LDL-C) by visit
Time Frame: Baseline, Day 90, Day 270 and Day 330
Population: Full Analysis Set (FAS) comprised all randomized participants. The number of participants analyzed corresponds to the number of subjects who had LDL-C values at baseline and Day 90, Day 270 and Day 330 respectively.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Inclisiran With Usual Care | Usual Care
Number analyzed (Participants) | 188 | 178
mg/dL
  Day 90 | -44.2 [-47.9 to -40.5] | -2.2 [-6.0 to 1.6]
  Day 270: number analyzed (Participants) | 175 | 158
  Day 270 | -34.6 [-39.2 to -30.1] | -3.8 [-8.6 to 1.0]
  Day 330: number analyzed (Participants) | 171 | 163
  Day 330 | -41.2 [-45.9 to -36.5] | -3.5 [-8.3 to 1.4]
Statistical Analysis 1: Comparison: Inclisiran With Usual Care vs Usual Care; Day 90; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS mean difference = -42.0, 95% CI 2-sided [-47.3 to -36.7]
Statistical Analysis 2: Comparison: Inclisiran With Usual Care vs Usual Care; Day 270; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS mean difference = -30.8, 95% CI 2-sided [-37.4 to -24.3]
Statistical Analysis 3: Comparison: Inclisiran With Usual Care vs Usual Care; Day 330; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS mean difference = -37.7, 95% CI 2-sided [-44.5 to -31.0]

4. Secondary Outcome: Average Percent Change From Baseline in LDL-C Levels
Description: Average percent change from baseline in low-density lipoprotein cholesterol (LDL-C) levels to each post-baseline visit
Time Frame: Baseline, from Day 90 to Day 330
Population: Full Analysis Set (FAS) comprised all randomized participants. The number of participants analyzed corresponds to the number of subjects who had at least one LDL-C change from baseline value available.
Measure: Least Squares Mean (95% Confidence Interval); unit: Average percent change in LDL-C
Arm/Group | Inclisiran With Usual Care | Usual Care
Number analyzed (Participants) | 194 | 184
Average percent change in LDL-C | -44.3 [-48.5 to -40.1] | 2.4 [-1.8 to 6.7]
Statistical Analysis 1: Comparison: Inclisiran With Usual Care vs Usual Care; Test type: Superiority; p < 0.001, ANCOVA; LS mean difference = -46.7, 95% CI 2-sided [-52.7 to -40.8]

5. Secondary Outcome: Average Absolute Change From Baseline in LDL-C Levels
Description: Average absolute change from baseline in low-density lipoprotein cholesterol (LDL-C) levels to each post-baseline visit
Time Frame: Baseline, From Day 90 to Day 330
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Inclisiran With Usual Care | Usual Care
Number analyzed (Participants) | 194 | 184
mg/dL | -40.0 [-43.6 to -36.4] | -2.7 [-6.4 to 1.0]
Statistical Analysis 1: Comparison: Inclisiran With Usual Care vs Usual Care; Test type: Superiority; p < 0.001, ANCOVA; LS mean difference = -37.3, 95% CI 2-sided [-42.4 to -32.2]

6. Secondary Outcome: Achieving ≥50% Reduction From Baseline in LDL-C
Description: Percentage of participants achieving ≥50% reduction from baseline in low-density lipoprotein cholesterol (LDL-C) at Day 330
Time Frame: Baseline, Day 330
Population: Full Analysis Set (FAS) comprised all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Inclisiran With Usual Care | Usual Care
Number analyzed (Participants) | 201 | 199
Percentage of participants | 45.3 [38.4 to 52.2] | 6.5 [3.1 to 10.0]
Statistical Analysis 1: Comparison: Inclisiran With Usual Care vs Usual Care; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 11.87, 95% CI 2-sided [6.33 to 22.25]

7. Secondary Outcome: Achieving LDL-C < 100 mg/dL and LDL-C < 55 mg/dL
Description: Percentage of participants achieving low-density lipoprotein cholesterol (LDL-C) <100 mg/dL (among the subset of participants with baseline LDL-C >= 100 mg/dL) and LDL-C < 55 mg/dL at Day 330
Time Frame: Day 330
Population: Full Analysis Set (FAS) comprised all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Inclisiran With Usual Care | Usual Care
Number analyzed (Participants) | 201 | 199
Percentage of participants
  Achieving LDL-C < 100 mg/dL: number analyzed (Participants) | 62 | 52
  Achieving LDL-C < 100 mg/dL | 75.8 [65.1 to 86.5] | 40.4 [27.0 to 53.7]
  Achieving LDL-C < 55 mg/dL | 54.2 [47.3 to 61.1] | 13.6 [8.8 to 18.3]
Statistical Analysis 1: Comparison: Inclisiran With Usual Care vs Usual Care; Achieving LDL-C < 100 mg/dL; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.38, 95% CI 2-sided [1.92 to 9.99]
Statistical Analysis 2: Comparison: Inclisiran With Usual Care vs Usual Care; Achieving LDL-C < 55 mg/dL; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 8.24, 95% CI 2-sided [4.97 to 13.65]

8. Secondary Outcome: Percent Change in Lipids and Other Lipoproteins From Baseline to Day 330
Description: Percent change in apolipoprotein B, very-low-density lipoprotein (VLDL), non-high-density lipoprotein cholesterol (non-HDL-C), total cholesterol, lipoprotein(a) (Lp[a]), HDL-C and triglycerides from baseline to Day 330
Time Frame: Baseline and Day 330
Population: Full Analysis Set (FAS) comprised all randomized participants. The number of participants analyzed corresponds to the number of subjects who had values at baseline and Day 330.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Inclisiran With Usual Care | Usual Care
Number analyzed (Participants) | 177 | 166
Percent change
  apolipoprotein B: number analyzed (Participants) | 168 | 164
  apolipoprotein B | -35.5 [-40.6 to -30.5] | 2.0 [-3.2 to 7.1]
  VLDL Cholesterol: number analyzed (Participants) | 175 | 165
  VLDL Cholesterol | 5.7 [-1.0 to 12.3] | 12.1 [5.2 to 18.9]
  non-HDL-Cholesterol: number analyzed (Participants) | 176 | 164
  non-HDL-Cholesterol | -35.2 [-39.6 to -30.8] | 2.5 [-2.0 to 7.1]
  Total Cholesterol | -21.4 [-24.7 to -18.1] | 4.1 [0.6 to 7.5]
  Lp[a]: number analyzed (Participants) | 160 | 158
  Lp[a] | -10.4 [-25.9 to 5.0] | 5.9 [-9.7 to 21.6]
  HDL-Cholesterol: number analyzed (Participants) | 176 | 164
  HDL-Cholesterol | 14.0 [10.8 to 17.3] | 10.6 [7.2 to 13.9]
  triglycerides | 7.3 [0.1 to 14.4] | 12.3 [4.9 to 19.6]
Statistical Analysis 1: Comparison: Inclisiran With Usual Care vs Usual Care; Apolipoprotein B; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS mean difference = -37.5, 95% CI 2-sided [-44.8 to -30.3]
Statistical Analysis 2: Comparison: Inclisiran With Usual Care vs Usual Care; VLDL Cholesterol; Test type: Superiority; p = 0.188, Mixed Models Analysis; LS mean difference = -6.4, 95% CI 2-sided [-16.0 to 3.1]
Statistical Analysis 3: Comparison: Inclisiran With Usual Care vs Usual Care; Non-HDL Cholesterol; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS mean difference = -37.7, 95% CI 2-sided [-44.0 to -31.4]
Statistical Analysis 4: Comparison: Inclisiran With Usual Care vs Usual Care; Total Cholesterol; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS mean difference = -25.5, 95% CI 2-sided [-30.2 to -20.7]
Statistical Analysis 5: Comparison: Inclisiran With Usual Care vs Usual Care; Lipoprotein(a); Test type: Superiority; p = 0.145, Mixed Models Analysis; LS mean difference = -16.4, 95% CI 2-sided [-38.4 to 5.7]
Statistical Analysis 6: Comparison: Inclisiran With Usual Care vs Usual Care; HDL Cholesterol; Test type: Superiority; p = 0.141, Mixed Models Analysis; LS mean difference = 3.5, 95% CI 2-sided [-1.2 to 8.1]
Statistical Analysis 7: Comparison: Inclisiran With Usual Care vs Usual Care; Triglycerides; Test type: Superiority; p = 0.339, Mixed Models Analysis; LS mean difference = -5.0, 95% CI 2-sided [-15.2 to 5.3]

9. Secondary Outcome: Absolute Change in Lipids and Other Lipoproteins From Baseline to Day 330
Description: Absolute change in apolipoprotein B, very-low-density lipoprotein (VLDL), non-high-density lipoprotein cholesterol (non-HDL-C), total cholesterol, HDL-C and triglycerides from baseline to Day 330
Time Frame: Baseline and Day 330
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Inclisiran With Usual Care | Usual Care
Number analyzed (Participants) | 177 | 166
mg/dL
  apolipoprotein B: number analyzed (Participants) | 168 | 164
  apolipoprotein B | -31.0 [-34.2 to -27.8] | -2.6 [-5.8 to 0.6]
  VLDL Cholesterol: number analyzed (Participants) | 175 | 165
  VLDL Cholesterol | -0.4 [-2.0 to 1.3] | 1.8 [0.0 to 3.5]
  non-HDL-Cholesterol: number analyzed (Participants) | 176 | 164
  non-HDL-Cholesterol | -41.4 [-46.5 to -36.3] | -1.3 [-6.5 to 4.0]
  total Cholesterol | -35.2 [-40.5 to -30.0] | 2.5 [-2.9 to 7.9]
  HDL-Cholesterol: number analyzed (Participants) | 176 | 164
  HDL-Cholesterol | 5.7 [4.3 to 7.1] | 3.8 [2.4 to 5.3]
  triglycerides | 1.1 [-8.7 to 10.8] | 9.8 [-0.3 to 19.9]
Statistical Analysis 1: Comparison: Inclisiran With Usual Care vs Usual Care; Apolipoprotein B; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS mean difference = -28.4, 95% CI 2-sided [-33.0 to -23.9]
Statistical Analysis 2: Comparison: Inclisiran With Usual Care vs Usual Care; VLDL Cholesterol; Test type: Superiority; p = 0.078, Mixed Models Analysis; LS mean difference = -2.1, 95% CI 2-sided [-4.5 to 0.2]
Statistical Analysis 3: Comparison: Inclisiran With Usual Care vs Usual Care; Non-HDL Cholesterol; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS mean difference = -40.1, 95% CI 2-sided [-47.5 to -32.8]
Statistical Analysis 4: Comparison: Inclisiran With Usual Care vs Usual Care; Total Cholesterol; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS mean difference = -37.7, 95% CI 2-sided [-45.3 to -30.2]
Statistical Analysis 5: Comparison: Inclisiran With Usual Care vs Usual Care; HDL Cholesterol; Test type: Superiority; p = 0.065, Mixed Models Analysis; LS mean difference = 1.9, 95% CI 2-sided [-0.1 to 3.8]
Statistical Analysis 6: Comparison: Inclisiran With Usual Care vs Usual Care; Triglycerides; Test type: Superiority; p = 0.222, Mixed Models Analysis; LS mean difference = -8.7, 95% CI 2-sided [-22.8 to 5.3]

10. Secondary Outcome: Absolute Change in Lp[a] From Baseline to Day 330
Description: Absolute change in lipoprotein(a) (Lp[a]) from baseline to Day 330
Time Frame: Baseline and Day 330
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Inclisiran With Usual Care | Usual Care
Number analyzed (Participants) | 160 | 158
nmol/L | -19.3 [-26.2 to -12.4] | -5.3 [-12.2 to 1.7]
Statistical Analysis 1: Comparison: Inclisiran With Usual Care vs Usual Care; Lipoprotein(a); Test type: Superiority; p = 0.005, Mixed Models Analysis; LS mean difference = -14.0, 95% CI 2-sided [-23.8 to -4.2]

11. Secondary Outcome: Intensity of Lipid Lowering Therapy
Description: Percentage of participants by intensity of lipid lowering therapy (dose decrease, increase or no change)
Time Frame: Baseline and Day 330
Population: Full Analysis Set (FAS) comprised all randomized participants. The number of participants analyzed corresponds to the number of subjects who had a record for Day 330 study visit date.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Inclisiran With Usual Care | Usual Care
Number analyzed (Participants) | 184 | 174
Percentage of participants
  Decrease in statin intensity | 9.8 [5.9 to 15.0] | 4.6 [2.0 to 8.9]
  No change in statin intensity | 89.1 [83.7 to 93.2] | 92.5 [87.6 to 96.0]
  Increase in statin intensity | 1.1 [0.1 to 3.9] | 2.9 [0.9 to 6.6]
Statistical Analysis 1: Comparison: Inclisiran With Usual Care vs Usual Care; Test type: Superiority; p = 0.031, proportional odds model; Odds Ratio (OR) = 0.43, 95% CI 2-sided [0.20 to 0.93]

12. Secondary Outcome: Proportion of Days Covered
Description: Total number of days on either statin, ezetimibe, or PCSK9 inhibiting monoclonal antibody therapies divided by total number of study days. If a participant did not take any of the 3 medications, then the total number of days was assumed to be zero.
Time Frame: Baseline through last date of participation, up to 330 Days
Population: Full Analysis Set (FAS) comprised all randomized participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: Proportion of days
Arm/Group | Inclisiran With Usual Care | Usual Care
Number analyzed (Participants) | 201 | 199
Proportion of days | 0.926 [0.900 to 0.953] | 0.965 [0.939 to 0.992]
Statistical Analysis 1: Comparison: Inclisiran With Usual Care vs Usual Care; Test type: Superiority; p = 0.043, ANCOVA; LS mean difference = -0.039, 95% CI 2-sided [-0.077 to -0.001]

13. Secondary Outcome: Discontinuation of Statin Therapy
Description: Percentage of participants discontinuing statin therapy. Discontinuation of statin therapy was defined as no statin use ≥ 30 days before the end-of-study visit.
  Participants for whom it could not be ascertained that they were on statin therapy at the end of study or who discontinued from the study early were assumed to have discontinued statin therapy.
Time Frame: Baseline and Day 330
Population: Full Analysis Set (FAS) comprised all randomized participants. Participants with Medical History of Statin Intolerance were excluded.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Inclisiran With Usual Care | Usual Care
Number analyzed (Participants) | 173 | 178
Percentage of participants | 14.5 [9.2 to 19.7] | 18.0 [12.3 to 23.6]
Statistical Analysis 1: Comparison: Inclisiran With Usual Care vs Usual Care; Test type: Superiority; p = 0.346, Regression, Logistic; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.43 to 1.35]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of 330 days.
Description: All safety analyses were conducted in the Safety Set.
Groups:
- Inclisiran + Usual Care: Inclisiran sodium 300 mg / 1.5 ml (equivalent to 284 mg of inclisiran) + usual care
Arm/Group | Inclisiran + Usual Care | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/203 | 2/197
Serious Adverse Events (participants affected / at risk) | 32/203 | 34/197
Other Adverse Events (participants affected / at risk) | 52/203 | 35/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inclisiran + Usual Care (N=203) | Usual Care (N=197)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 8 | 6
Angina pectoris (Cardiac disorders) | 2 | 2
Angina unstable (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Bundle branch block left (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 2
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 2 | 0
Cardiac perfusion defect (Cardiac disorders) | 1 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 2 | 1
Heart failure with preserved ejection fraction (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Blindness unilateral (Eye disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Muscle abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Varicella zoster virus infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Dysarthria (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 2
Lethargy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Tremor (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal artery thrombosis (Renal and urinary disorders) | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypertensive emergency (Vascular disorders) | 1 | 0
Hypertensive urgency (Vascular disorders) | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Inclisiran + Usual Care (N=203) | Usual Care (N=197)
Angina pectoris (Cardiac disorders) | 7 | 3
Injection site pain (General disorders) | 10 | 0
Non-cardiac chest pain (General disorders) | 8 | 10
COVID-19 (Infections and infestations) | 10 | 9
Upper respiratory tract infection (Infections and infestations) | 6 | 6
Blood creatine phosphokinase increased (Investigations) | 5 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 3
Dizziness (Nervous system disorders) | 6 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/34/NCT04873934/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-29): https://cdn.clinicaltrials.gov/large-docs/34/NCT04873934/SAP_001.pdf